CLINICAL TRIAL: NCT07225179
Title: Bolster-NC: A Pilot Study of the Bolster mHealth Intervention Within Early Psychosis Program Outreach in North Carolina
Brief Title: mHealth for Early Psychosis Caregivers in Statewide Program Outreach
Acronym: Bolster-NC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: North Carolina Department of Health and Human Services (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-1793
Record Dates: First submitted 2025-11-03; First posted 2025-11-06 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Caregiver; Caregiver Distress; Caregiver to a Young Adult With Early Psychosis; Family Caregivers
Keywords: Caregiver; Caregiver Support

STUDY DESIGN:
Intervention Model Description: Single group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bolster (Experimental): Participants will be provided access to the Bolster smartphone application designed to support caregivers of young adults with early psychosis. They will also have access to the research team by phone for technical troubleshooting and support as necessary.
  Interventions: Behavioral: Bolster

INTERVENTIONS:
Behavioral: Bolster — Bolster is a native mobile app that provides on-demand content to caregivers of young adults with early psychosis to support their caregiving skills and knowledge of psychosis. Participants will also have access to a member of the study team for technical troubleshooting and support as necessary.

SUMMARY:
The purpose of this study is to pilot the delivery of an mHealth intervention for caregivers to young people with early psychosis within a network of early psychosis intervention programs in the state of North Carolina. The investigators will examine the feasibility of recruitment through program outreach, develop North Carolina specific outreach resources to be used with the mHealth intervention and evaluate the effectiveness of this intervention for reducing caregiver psychological morbidity and improving family communication. The investigators will also collect pilot data to inform recruitment and development of implementation strategies for delivering Bolster within a statewide early psychosis network.

DETAILED DESCRIPTION:
The team aims to pilot test the delivery of an mHealth intervention for caregivers to young people with early psychosis within a network of early psychosis intervention programs in the state of North Carolina. This will involve (1) examining the feasibility of recruitment through program outreach, (2) developing and optimizing state-specific outreach resources and recruitment approaches to be implemented for this mHealth intervention, and (3) evaluating the effectiveness of this intervention in reducing caregiver psychological morbidity and improving family communication. Participants will be caregivers to young people experiencing early psychosis within the state of North Carolina. Remote recruitment resources will be developed and distributed through the EPI-NC outreach program (i.e. network of UNC-based early psychosis clinicians and stakeholders aiming to raise awareness of early psychosis and specialty programs). Recruited participants will complete baseline measures and be given access to the Bolster mHealth intervention, which provides self-guided psychoeducation and communication coaching for early psychosis caregivers. The investigators will collect baseline and post-test data and evaluate within-subjects changes in proposed targets and outcomes including primary outcomes of caregiver psychological morbidity and family communication.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* North Carolina resident
* Caregiver to a young adult with early psychosis, wherein early psychosis is defined as: (1) Being between the ages of 15 and 30, and (2) Within the past five years, the young adult first experienced hallmark symptoms: (2A) Presence of psychotic symptoms represented by one or more of hallucinations, delusions, marked thought disorder, psychomotor disorder or bizarre behavior, as well as (2B) Definite change of personality or behavior manifesting as two or more of the following: serious deterioration of function, marked social withdrawal, persistent self-neglect, episodic marked anxiety.
* A positive screen according to the Caregiver Prime Screen - Revised (endorsed two or more responses of five or six ("somewhat"/"definitely" agree)
* Own an Apple iPhone
* Have access to the internet (e.g., via WiFi or data plan)
* Self-identify as a caregiver of the affected person
* Are proficient in English to the degree necessary to complete study assessments and engage meaningfully in the intervention

Exclusion Criteria:

* Participant failed to demonstrate understanding of study details in comprehension screening process.
* Previous enrollment in a study involving Bolster.
* Activity on screening questionnaires that indicates suspicious or dishonest participation such that the participant is likely to be a "malicious actor" or "gamer" (i.e. an individual that attempts to enroll in online research studies solely for compensation with dishonest or illegitimate responses to study questionnaires)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Change in family communication / expressed emotion | Baseline, 12 weeks
  Family communication will be assessed with the Family Questionnaire (FQ). The FQ is a 20-item self-report assessment of criticism and emotional expression in interactions with family members toward patients with mental illness. Each item is rated on a 4-point scale (1 = never/very rarely; 4 = very often). The FQ is scored by summing individual items with higher scores indicating greater levels of expressed emotion. As a primary outcome, the investigators will examine the combined total of emotional overinvolvement and critical comments; scores range from 20 to 80 with higher scores indicating greater expressed emotion.
Change in caregiver psychological morbidity | Baseline, 12 Weeks
  Caregiver psychological morbidity will be assessed with General Health Questionnaire (GHQ), a 12-item questionnaire assessing general psychological morbidity. Respondents indicate agreement on a four-point scale (0 = Not at all; 3 = More than usual) and total scores ranging from 0 to 36 with higher scores indicating more severe psychological morbidity.

SECONDARY OUTCOMES:
Change in illness knowledge | Baseline, 12 weeks
  Caregiver perception of illness knowledge will be assessed using the Illness Perception Questionnaire for Schizophrenia Relatives (IPQ), a self-report scale of caregivers' beliefs about the severity, prognosis, and responsiveness to treatment of mental illness. The investigators will examine the illness coherence scale as a measure of self-perceived knowledge/understanding of psychosis, a 5-item score (ranging from 5 to 25) denoting the extent to which one feels that one has a coherent understanding of the mental health problem. Higher scores suggest higher self-perceived knowledge/understanding of psychosis.
Change in emotional distress about illness | Baseline, 12 weeks
  Illness appraisals will be assessed with the Illness Perception Questionnaire for Schizophrenia Relatives (IPQSR), a self-report scale of caregivers' beliefs about the severity, prognosis, and responsiveness to treatment of mental illnesses. Each item is rated on a 5-point scale (1 = strongly disagree; 5 = strongly agree), and totals are scored by summing individual items. For the emotional distress score, the investigators are examining the emotional representation scale, a 9-item scale with scores ranging from 9 to 45, with higher scores indicating greater emotional distress.
Change in coping self-efficacy | Baseline, 12 weeks
  Caregiver coping self-efficacy will be assessed with the Coping Self-Efficacy Scale, a 26-item self-report questionnaire measuring the perceived ability of coping with various life challenges. Responses are rated on a 0 to 10 scale, and scores range from 0 to 260, with higher scores denoting a greater sense of self-efficacy in coping.
Change in appraisals of caregiving experiences | Baseline, 12 weeks
  Appraisals of caregiving experiences will be assessed with the Brief Experience of Caregiving Inventory (BECI). The BECI is a 19-item assessment of the impact of caregiving on the individual's life, both in negative and positive ways. The items are rated on a 5-point Likert scale (never to nearly always), and scores range from 0 to 76, with a higher score denoting more negative appraisals of one's caregiving experience.

CONTACTS AND LOCATIONS:
Overall Officials: Ben Buck, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC Department of Psychiatry, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 12 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Time Frame: Beginning 12 and continuing for 36 months following publication
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.